CLINICAL TRIAL: NCT02215317
Title: Impact of Obstructive Sleep Apnea on Cardiovascular Outcomes in Patients Treated With Percutaneous Coronary Intervention
Brief Title: Sleep and Stent Study: a Multicentre, Prospective Study
Status: Completed | Type: Observational
Sponsor: National University of Singapore (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Chi-Hang Lee, Associate Professor, National University of Singapore
Other Study IDs: SSS
Record Dates: First submitted 2014-08-08; First posted 2014-08-13 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep Apnea; Stent; Coronary Artery Disease; Percutaneous Coronary Intervention
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- OSA group: Patients found to have OSA based on an overnight sleep study
- Non-OSA group: Patients found not to have OSA based on an overnight sleep study

SUMMARY:
Elucidating the effects of obstructive sleep apnea (OSA) on cardiovascular outcomes is crucial in risk assessments and therapeutic recommendations for affected individuals. The Sleep and Stent Study is a multi-center observational study investigating the relationships between OSA and cardiovascular outcomes in patients treated with percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Preliminary data suggest that OSA may lead to adverse cardiovascular outcomes after PCI. However, existing data were generated from small-scale, single-center studies. Therefore, in the Sleep and Stent Study, the investigators aim to conduct a large-scale multi-national cohort study to determine the association between OSA and the incidence of adverse cardiovascular outcomes over a long-term follow-up period. The investigators hypothesize that OSA is an independent risk factor for the development of major adverse cardiovascular and cerebrovascular events (MACCEs) in coronary artery disease patients treated with PCI. Results from the Sleep and Stent Study will advance the fundamental understanding of the burden and prognostic implications of OSA in patients undergoing PCI for coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and < 80 years old
* Successful PCI to at least one of the epicardial coronary arteries

Exclusion Criteria:

* Known OSA on CPAP treatment
* Intubation for mechanical ventilation
* Intra-aortic balloon pump or other hemodynamic support device
* Sedation or other muscle relaxant given before overnight sleep study
* Perceived high risk of malignant ventricular arrhythmia
* Cardiogenic shock with systolic blood pressure <90 mmHg
* Clinical heart failure requiring oxygen supplementation
* Pregnancy
* History of malignancy (except non-melanoma skin cancer, cervical in-situ carcinoma, breast ductal carcinoma in situ or stage 1 prostate carcinoma)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, observational multi-national cohort study of patients undergoing PCI for coronary artery disease. Adult patients undergoing clinically indicated PCI for coronary artery disease will be enrolled in the Sleep and Stent Study.
Sampling Method: Non-Probability Sample
Enrollment: 1815 (Actual)
Dates: Start 2011-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Major Adverse Cardiac and Cerebrovascular events (MACCE) | Two years
  Cardiovascular Death, Myocardial Infarction, Stroke/TIA, Unplanned revascularization

SECONDARY OUTCOMES:
Number of Participants with Adverse Events other than MACCE | Two years
  All-cause mortality, Target vessel revascularization, Stent thrombosis, Hospitalization for heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hang Lee, MD, Principal Investigator — National University Heart Centre, Singapore
Locations (1):
- Venesa Loh, Singapore, Singapore

REFERENCES:
- [Background] Loo G, Koo CY, Zhang J, Li R, Sethi R, Ong TH, Tai BC, Lee CH. Impact of obstructive sleep apnea on cardiovascular outcomes in patients treated with percutaneous coronary intervention: rationale and design of the sleep and stent study. Clin Cardiol. 2014 May;37(5):261-9. doi: 10.1002/clc.22261. PMID 24945037